CLINICAL TRIAL: NCT01025388
Title: Centralized Pan-Middle East Survey on the Undertreatment of Hypercholesterolemia
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: ClinArt Company & Signen Clinical Discoveries (Unknown)
Responsible Party: Sponsor
Other Study IDs: NIS-SA-CRE-2009/1
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2011-05

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; The study is focusing on the undertreatment of hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the NCEP ATP III/updated 2004 NCEP ATP III guidelines, overall and by country, in the following sub-populations:

* Primary/secondary prevention patients.
* Patients with metabolic syndrome (according to NCEP III definition).

In addition, the purpose is to establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the Third Joint European Task Force guidelines/national guidelines, in the survey population and in the following sub-populations:

* Primary/secondary prevention patients.
* Patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* On lipid-lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks. ·
* Subject must sign informed consent

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject who visits the primary care clinics, cardiology clinics and internal medicine clinics, and who fulfil the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 4053 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the NCEP ATP III / updated 2004 NCEP ATP III guidelines, overall and by country. | 6 months- One visit only, no follow up visits.

SECONDARY OUTCOMES:
The proportion of patients reaching the LDL-C goals according to the NCEP ATP III/updated 2004 NCEP ATP III in the following sub-populations - Primary/secondary prevention patients - Patients with metabolic syndrome (according to NCEP III definition). | 6 months - One visit only, no follow up visits.
The proportion of patients reaching the LDL-C goals according to the Third Joint European Task Force guidelines / national guidelines, in the following sub-populations:-Primary/secondary prevention patients -Patients with metabolic syndrome. | 6 months- One visit only, no follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Mohammed Arafah, Study Chair — King Khalid University Hospital; Dr. Shorook Alherz, Principal Investigator — King Fahad National Guard Hospital; Dr. Khalid Alnemer, Principal Investigator — Security Forces Hospital; Dr. Hossam Alghetany, Principal Investigator — Soliman Fakieh Hospital; Dr. Othman Metwally, Principal Investigator — King Fahad General Hospital; Dr. Akram Alkhadra, Principal Investigator — King Fahad University Hospital; Dr. Faisal Alanizi, Principal Investigator — Ministry of Health, Saudi Arabia
Locations (5):
- Saudi Arabia (5):
  - Research Site, Riyadh, Central
  - Research Site, Dammam, Eastern Province
  - Research Site, Aljouf, North
  - Research Site, Jeddah, Western
  - Research Site, Makah, Western